CLINICAL TRIAL: NCT07329231
Title: Quinoa Improves Glycolipid Metabolism and Glucose Fluctuation Based on β-Cell Function in Early-stage Type 2 Diabetes
Acronym: QIGMAGFBOβFIET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, kuanxiao Tang, chief physician, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-2019(ZM)-062
Record Dates: First submitted 2025-06-01; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Diabetes Mellitus; Quinoa Dietary Intervention; Glycaemic Fluctuations; Glycolipid metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the quinoa diet (QD) group (Experimental): The QD group replaced part of their staple foods with quinoa noodles, mixed flour, and biscuits. The intervention lasted for 14 weeks. Regular monitoring of indicators such as blood sugar, blood lipids, insulin resistance (HOMA-IR), and β-cell function (HOMA-β) was conducted, and the use of medications was recorded.
  Interventions: Dietary Supplement: Quinoa-based foods
- the regular diet (RD) group (No Intervention)

INTERVENTIONS:
Dietary Supplement: Quinoa-based foods — Quinoa-based foods included three varieties: quinoa noodles (80 g per bag; the ingredients included quinoa powder, red bean powder, black wheat powder, black mung bean powder, and edible salt, with quinoa powder comprising 15% of the total produced by Shandong Tangren Duoyi Biotechnology Company), blended powder (15 g per bag; the ingredients included quinoa, rye wheat, black mung beans, adzuki beans, black sesame seeds, chickpeas, konjac flour, and mogroside, with quinoa flour comprising 20% of the total produced by Shandong Tangren Duoyi Biotechnology Company), and cookies (24 g per bag; quinoa, rye, adzuki beans, black sesame seeds, vegetable oil, and salt, with quinoa comprising 20% of the total produced by Shandong Tangren Duoyi Biotechnology Company). These products serve as substitutes for the common starchy staples, soups, porridge, and snacks typically consumed by T2DM patients. This substitution did not alter patients' daily eating habits; rather, it simply replaced tradition
  Arms: the quinoa diet (QD) group

SUMMARY:
The goal of this clinical trial is to explore whether quinoa diet can improve glycolipid metabolism and glucose fluctuations in patients with early-stage type 2 diabetes mellitus (T2DM) and observe its impact on islet β-cell function and insulin resistance in patients with early-stage T2DM (diagnosed according to the 1999 WHO criteria, disease duration <5 years, HbA1c 6.5%-10%, no history of insulin therapy, aged 20-70 years).

The main question it aims to answer is:

Can quinoa diet reduce blood glucose (fasting blood glucose, postprandial blood glucose, glycosylated hemoglobin), improve lipid metabolism (cholesterol, triglycerides), and stabilize glucose fluctuations (time in range, time above range) in patients with early-stage T2DM? Does quinoa diet improve islet β-cell function (HOMA-β) and insulin resistance (HOMA-IR), and reduce the need for oral hypoglycemic medications? Comparison group: Researchers will compare the quinoa diet (QD) group (replacing traditional starchy foods with quinoa products) vs. the regular diet (RD) group (conventional diet) to see if quinoa diet demonstrates better metabolic improvement and medication reduction effects.

Participants will:

Be randomly assigned to the QD group or RD group. Undergo oral glucose tolerance tests (OGTTs) and continuous glucose monitoring (cGMS) at baseline and after the intervention.

The QD group will consume quinoa-based foods (noodles, blended powder, cookies) as substitutes for staple foods, beverages, and snacks for 14 weeks, documenting daily intake in a record book.

Both groups will receive standardized dietary and exercise education, with monthly follow-ups for food distribution and data collection.

ELIGIBILITY:
Inclusion Criteria:

patients diagnosed according to the 1999 WHO diagnostic criteria for T2DM with a duration of less than 5 years HbA1c levels between 6.5% and 10% no history of insulin therapy age between 20 and 70 years. Exclusion Criteria： acute complications of diabetes, such as diabetic ketoacidosis severe acute or chronic conditions affecting the liver, kidneys, heart, cerebrovascular system, gastrointestinal tract, or acute infectious diseases pregnancy or plans for pregnancy soon allergies to quinoa or bean products participation in other dietary interventions or drug clinical trials within the past three months gastrointestinal diseases within two weeks prior to enrolment.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Glucose variability (MAGE) assessed by continuous glucose monitoring | From registration to the end of the 14-week treatment
  Change from baseline to week 14 in Mean Amplitude of Glycemic Excursions (MAGE) calculated from 72-hour continuous glucose monitoring data.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-06-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT07329231/ICF_000.pdf